CLINICAL TRIAL: NCT01148381
Title: Characterization of Phenotypic and Genotypic Regressors
Brief Title: Characterization of Phenotypic and Genotypic Regressors for Imaging
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910457; 10-DA-N457
Record Dates: First submitted 2010-06-19; First posted 2010-06-22 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: Healthy Volunteers; Substance Use Disorders
Keywords: Genotype; Phenotype; Characterization; fMRI; Natural History
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- controls: healthy non-smoking, participants with no substance use disorders
- psychiatric disorders: individuals with other psychiatric disorders
- smokers: healthy individuals with nicotine use disorder
- substance use disorders: healthy individuals with other substance use disorders
- treatment seeking individuals: treatment seeking individuals with substance use disorders

SUMMARY:
The influence of genes on addictive and neuropsychiatric disorders is complex, especially given that multiple genes likely influence certain behaviors that are correlated with addiction. Researchers are interested in looking at the genetic information of individuals who are enrolled on National Institute for Drug Abuse studies to investigate specific genetic variants that may be related to substance abuse. Researchers will study the effects of genes on several aspects of thinking such as attention, memory, decision making, problem solving, learning, and emotional feelings, and investigate the ways in which genetic information affects addictive behaviors and substance abuse. In addition, researchers will study how genes may explain differences in imaging data in substance users.

Objectives:

- To collect genetic information for research on genetic aspects of addiction and substance abuse.

Eligibility:

* Adults age 18 or older

  * (1) healthy, non-drug-using nonsmokers,
  * (2) healthy smokers,
  * (3) healthy individuals dependent on other commonly abused drugs, and
  * (4) individuals with other psychiatric disorders.
* Participants must be enrolled in another National Institute on Drug Abuse, Intramural Research Program imaging protocol.

Design:

* This study involves one to two visits to National Institute on Drug Abuse, Intramural Research Program that may be separate from the participant's current research protocol study visits or on the same day as those visits.
* Participants will provide a blood sample and complete questionnaires about mood, memory, and learning.
* Participants may also be asked to do a few tasks, such as playing computer games involving coin tosses and money management, or responding to questions on a computer screen.

DETAILED DESCRIPTION:
Objective: To determine genetic variants as well as behavioral measures across different study group populations. Results of these will be used as regressors to help explain inter-individual differences in data collected across IRP protocols.

Study Population: The study population will include 1) healthy non-smoking, participants with no substance use disorders 2) healthy individuals with nicotine use disorder 3) healthy individuals with other substance use disorders 4) individuals with other psychiatric disorders and 5) treatment-seeking individuals with substance use disorders. Participants must be under evaluation for another NIDA-IRP protocol, generally healthy, and age 18 or older.

Design: The main study will require approximately 5-8 hours. Main study procedures may be done in 1 visit or multiple visits, and may be done in conjunction with another NIDA-IRP study. After being consented into the main study, the participant will be asked to submit a blood sample, an MRI scan, complete various questionnaires, characterization instruments and several behavioral tasks. Blood will only be drawn once, provided there are no technical problems (such as sample damage during collection, preparation, shipping or assay) requiring a repeat draw. If participants enroll in other NIDA-IRP imaging protocols, they will be asked to repeat a few of the time- sensitive questionnaires in this protocol during the MRI visits of the other protocols. Data acquired in this protocol will be compared to data acquired in other NIDA-IRP protocols.

An arm of this protocol will be used to pilot test a phenotyping battery developed by the NIDA CTN. This battery overlaps with several of the assessments in the main protocol. Participants in the NIDA CTN pilot study who also meet criteria for the main study may participate in the main study as well. The CTN Pilot procedures require approximately 4-6 hours to complete.

Outcome Measures: The primary outcome measures in this study are the genetic, behavioral and phenotypic factors that are related to addiction. Secondary outcome measures are to compare the genetic, behavioral and phenotypic factors to imaging and behavioral data acquired across other IRP protocols.

ELIGIBILITY:
* INCLUSION CRITERIA: Main Study

All participants must be:

-under evaluation for or enrolled in another NIDA-IRP study. Justification: This protocol is primarily meant to gather uniform characterization data on IRP participants although the data is useful regardless of participation in other protocols.

->= 18 years of age. Justification: The majority of NIDA-IRP studies only include adults, as such, we will only include adults in this study for now.

EXCLUSION CRITERIA: Main Study.

* History of neurological illnesses that per the study clinicians would be significant enough to impair ability to tolerate the procedure or alter neuronal activity, including but not limited to CVA, CNS tumor, head trauma with significant sequelae, Multiple Sclerosis or other demyelinating diseases, epilepsy, movement disorders, or migraine in treatment. Assessment tool: History and physical (H&P). Rationale: Neurological illnesses may impair ability to tolerate the procedures and alter neuronal activity, adding noise to the data.
* Cognitive impairment (unless this population of subjects is included in another IRP protocol for which the subject is also under consideration). Assessment tool: self-report during H&P of special education classes, history of specific learning disability or mental retardation. A validated IQ test such as the Shipley-2 may also be administered. Rationale: Cognitive impairment may impair ability to tolerate the procedures and alter neuronal activity, adding noise to the data.
* Current major mood, anxiety or psychotic disorder (unless this population of subjects is included in another IRP protocol for which the subject is also under consideration). Assessment tool: self-report, H&P, a structured or semi-structured psychiatric interview such as the computerized SCID with follow up clinical interview (or full interviewer-administered). Rationale: Current major mood or psychotic disorders may impair ability to tolerate the procedures and alter neuronal activity, adding noise to the data.
* Pregnancy. Assessment tool: Urine pregnancy test. Rationale: fMRI is not accepted as a safe procedure purely for research purposes during pregnancy.
* HIV -positive individuals. Assessment tool: oral HIV test with serum confirmation of positive results. Rationale: potential liver/metabolic/vascular disease can interfere with the physiological transduction mechanisms for fMRI (i.e. making the measurement unreliable).
* Unable to undergo MRI scanning due to possible pregnancy, metallic devices in the body, claustrophobia or body morphometry.
* Currently using respiratory, cardiovascular or anticonvulsant medications that may interfere with the BOLD MRI signal.
* Non-English speaking. Assessment tool(s): self-report. Rationale: To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify given the small sample size for each experiment. Additionally, the data integrity of some of the cognitive tasks and standardized questionnaires used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing study procedures. The inability to effectively communicate safety procedures in a language other than English could compromise the safety of non-English speaking participants.
* Other health conditions that would impact safety of participation or scientific integrity of data collection.

Inclusion criteria: NIDA CTN Pilot Study

All participants must:

1. Either have a current DSM-5 diagnosis for at least one of the following substance use disorders: nicotine, cocaine, marijuana, opiate; or 2) no current DSM-5 substance use disorder (control participants). Justification: These criteria are consistent with the scope of this study to pilot this battery of tests for future use in similar populations enrolled in the NIDA CTN studies.
2. Be >= 18 years of age. Justification: The NIDA CTN will use this battery in adults.

Exclusion criteria: NIDA CTN Pilot Study

1. A DSM-5 major psychiatric diagnoses unrelated to a substance use disorder including but not limited to bipolar disorder and schizophrenia. Diagnoses secondary to substance use disorder will be allowable providing the participant's symptoms do not interfere with the ability to complete assessments. Assessment tool: self-report, H&P, structured or semi-structured psychiatric interview.

   Rationale: Current major mood or psychotic disorders may impair ability to complete the assessments and would add unnecessary noise to the data.
2. Cognitive impairment. Assessment tool: self-report during H&P of special education classes, history of specific learning disability or mental retardation. A validated IQ test such as the Shipley-2 may also be administered. Rationale: Cognitive impairment may impair ability to complete the assessments and would add unnecessary noise to the data.
3. Non-English speaking. Assessment tool(s): self-report. Rationale: To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify given the small sample size for each experiment. Additionally, the data integrity of some of the cognitive tasks and standardized questionnaires used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing study procedures. The inability to effectively communicate safety procedures in a language other than English could compromise the safety of non-English speaking participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the main study, subjects will be recruited from the pool of subjects who are being considered for other NIDA-IRP protocols. Therefore, participant distribution in the main study will reflect that specified in other NIDA-IRP protocols. No preferences in participant recruitment will be made on the basis of sex, race, or ethnic background. In both the main study and the CTN pilot, efforts will be made to include ethnic minorities in proportion to their presence in the Baltimore City area, which is where the majority of our subjects reside.
Sampling Method: Non-Probability Sample
Enrollment: 847 (Actual)
Dates: Start 2010-11-18 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are the genetic, behavioral and phenotypic factors that are related to addiction. | each visit
  To determine whether genetic polymorphisms, phenotypic measures and behavioral characterization instruments can explain variance in structural and functional imaging data and in behavioral outcome measures such as treatment outcome or substance use trajectories or patterns as collected under other NIDA IRP protocols and clinical trials conducted in the NIDA CTN.

SECONDARY OUTCOMES:
Secondary outcome measures are to compare the genetic, behavioral and phenotypic factors to imaging and behavioral data acquired across other IRP protocols. | each visit
  To compare the genetic, behavioral and phenotypic factors to imaging and behavioral data acquired across other IRP protocols

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Janes, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided